CLINICAL TRIAL: NCT02954744
Title: Therapeutic Efficacy of High-intensity Focused Ultrasound in the Treatment of Uterine Fibroid
Brief Title: High-intensity Focused Ultrasound in Treatment of Uterine Fibroid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Vincent YT Cheung, Dr, Queen Mary Hospital, Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW11-204
Record Dates: First submitted 2016-10-20; First posted 2016-11-03 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Fibroids
Keywords: uterine fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): HIFU treatment
  Interventions: Procedure: HIFU treatment

INTERVENTIONS:
Procedure: HIFU treatment — High intensity focused ultrasound

SUMMARY:
Uterine fibroids are common uterine benign neoplasm. They can cause abnormal menstrual bleeding, pelvic discomfort and urinary frequency. Although surgical intervention is the definitive treatment, some women prefer to have their uterus preserved. High-intensity focused ultrasound (HIFU) therapy is receiving increasing interest in the management of uterine fibroids by inducing focal thermocoagulation of the fibroids. Results obtained by various research groups have shown that HIFU treatment is safe, effective and is highly acceptable to patients. The main objective of this study is to evaluate the therapeutic efficacy of HIFU in the treatment of uterine fibroids.

In this proposed study, 20 patients who have symptomatic uterine fibroids who meet the study inclusion criteria will be invited to participate in the study which involves the use of HIFU in the management of the fibroid. Background information of the patients such as age, body mass index, hormonal (pre- or postmenopausal) status and the presence of chronic medical disease will be collected. Subjects will also be asked to complete an eight-item section of a Uterine Fibroid Symptom and Quality Of Life Questionnaire (UFS-QOL) which evaluate the effect of the fibroid on the quality of life of women.

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years old, with no future childbearing plans
* Age >30 years old, who has tubal sterilization
* Significant fibroids symptoms
* Clinical uterine size less than 20 weeks gestation
* Dominant fibroid less than 10 cm in diameter without areas of necrosis as judged by contrast MRI
* No laparotomy scars
* Women should be able to give consent

Exclusion Criteria:

* Other pelvic or uncontrolled systemic diseases
* Confirmed or suspected pregnancy
* Patients who are contraindicated for MRI examination
* Patients with thick abdominal wall (>5 cm, as measured by MRI)
* Presence or history of acute pelvic inflammatory disease
* History of lower abdominal surgery, known severe pelvic endometriosis and/ or extensive pelvic adhesion
* Cervical fibroids, subserous or submucous fibroids with pedicle, <3.5 cm posterior wall fibroid, fibroids suspicious of malignancy (rapidly growing)

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2017-08 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of HIFU in reducing the size of the uterine fibroids by sonographic measurements | The changes from baseline to post12-month treatment will be captured
  By sonographic measurements at baseline, post 1-month, post 3-month, and post 12-month, the size of the uterine fibroids will be evaluated by physicians

SECONDARY OUTCOMES:
Patient satisfaction score after HIFU treatment of uterine fibroid | Up to 12 months
  Patients will be asked to give the satisfaction score (0= not satisfactory, 5= very satisfactory) at each follow up (i.e. post treatment 1 months, 3 months, 6 months and 12 months)
Change of perceived symptoms after HIFU treatment by using the Uterine Fibroid Symptoms Quality Of Life Questionnaire (UFS_QOL) | Up to 12 months
  By using the Uterine Fibroid Symptoms Quality Of Life Questionnaire (UFS_QOL) at each follow up (i.e. from baseline to post 1- month, post 1-month to post 3-month, post 3-month to post 6-month, post 6-month to post 12-month treatment will be captured).
Risks and adverse effects of HIFU in the treatment of uterine fibroid | Up to 12 months
  Patient will be evaluated for abnormal laboratory values and/or adverse events that are related to treatment at each follow up (i.e. post treatment 1 months, 3 months, 6 months and 12 months)
Subsequent management after HIFU treatment of uterine fibroid | Up to 12 months
  By physician's judgment at each follow up (i.e. at post treatment 1 months, 3 months, 6 months and 12 months), the need for subsequent additional treatments (such as hysterectomy, uterine artery embolization, or any type of hormonal treatment) will be evaluated.
Efficacy of HIFU in reducing the size of the uterine fibroids by MRI measurements | The changes from baseline to post 6-month treatment will be captured
  By MRI measurements at baseline, post 6-month, the size of the uterine fibroids will be evaluated by physicians

CONTACTS AND LOCATIONS:
Overall Officials: Vincent, YT Cheung, MBBS, FRCOG, Principal Investigator — Queen Mary Hospital, Hong Kong